CLINICAL TRIAL: NCT04077450
Title: Effectiveness of Heart-focused Breathing on Reducing Burden in Alzheimer's Caregivers: An Online Randomized Pilot Study
Brief Title: Heart-Focused Breathing in Alzheimer's Disease Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed the direction and aims of the study
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009353
Record Dates: First submitted 2019-08-02; First posted 2019-09-04 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Burnout, Caregiver; Quality of Life
Keywords: Stress; Caregiver Burden; Alzheimer's Disease Caregiver; Informal Caregiver; Anxiety; Heart-Focused Breathing
MeSH Terms: conditions — Caregiver Burden; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which participants will be randomized into (a) the modified waitlist-control arm or (b) the intervention arm.
Who Masked: Participant
Masking Description: Only participants will be blinded as to which study arm he or she was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Waitlist Control Arm (No Intervention): Participants will complete the following components of baseline (T1) data collection: demographics, questionnaire, heart rate variability assessment. Two weeks later, participants will be asked to complete post-intervention data collection (T2), which consists of a questionnaire and heart rate variability assessment. After the completion of data collection, participants will be offered the online heart-focused breathing intervention.
- Intervention Arm (Experimental): Participants will complete the following components of baseline (T1) data collection: demographics, questionnaire, heart rate variability assessment. These participants will receive an online heart-focused breathing intervention. Participants will be asked to practice their breathing skills while monitoring their heart rate variability using the Welltory app on their smart device for the following two weeks. Participants will be instructed to maintain a log to record the date and time of each practice session. Research staff will make biweekly reminder calls to participants. After the two-week period, participants will complete post-intervention data collection (T2), which includes a questionnaire and HRV assessment.
  Interventions: Behavioral: Online Heart-Focused Breathing Intervention

INTERVENTIONS:
Behavioral: Online Heart-Focused Breathing Intervention — Participants will receive an online standardized HeartMath© heart-focused breathing intervention.
  Arms: Intervention Arm

SUMMARY:
This research study will explore the effects of an online heart-focused breathing intervention on 20 informal caregivers of patients with Alzheimer's Disease (AD) over a period of two weeks.

DETAILED DESCRIPTION:
Informal caregivers are often live-in, unpaid spouses, relatives, partners, or friends that help with a loved one's activities of daily living. As a result of caring for a person with Alzheimer's Disease (AD), many informal caregivers experience caregiver burden. The demanding physical, emotional, and financial responsibilities to care for an AD patient can be detrimental to the caregiver's health.

A group of 20 men and women who consider themselves the primary caregiver of a person with AD will be recruited and enrolled into the study. Participants will be randomized into one of two study arms, (a) the modified-waitlist control arm or (b) the intervention arm. The study will explore the effects of an online heart-focused breathing intervention on heart rate variability (measured by the Welltory app on their smart device), perceived burden, stress, and quality of life in the intervention arm over a two-week period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Live-in and unpaid informal caregiver to a loved one with Alzheimer's Disease
* Provides care or supervision for at least 4 hours per day for more than 6 months
* Experiencing stress

Exclusion Criteria:

* Caregivers who report a low risk assessment score and/or report a medically diagnosed arrhythmia or have a pacemaker will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden | 2 weeks
  Caregiver Burden will be measured by the Zarit Burden Interview short version (12 items, 5-point Likert scale; 0= never, 4= nearly always). Score range= 0 to 48. A score of 17 or higher indicates a high level of burden.

SECONDARY OUTCOMES:
Life Quality | 2 weeks
  Quality of Life will be measured by the Arizona Integrative Outcomes Scale (AIOS) (2-items, visual analogue scale; 0 millimeters= worst you have ever been, 100 millimeters= best you have ever been). Score range= 0 to 200. The AIOS asks participants to reflect on their sense of well-being over the past 24 hours and over the past month.
Perceived Stress | 2 weeks
  Perceived Stress will be measured by the Perceived Stress Scale (PSS) (10 items, 5-point Likert scale; 0= never, 4= very often). Score range= 0 to 40. The PSS has a general score by combining all item scores and reverse scoring items 4, 5, 7, and 8. The PSS has two subscales, one for perceived distress (items 1, 2, 3, 6, 9, 10) and one for perceived coping (4, 5, 7, 8). A higher general score is associated with a higher level of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No